CLINICAL TRIAL: NCT06982924
Title: A Prospective, Controlled Phase II Clinical Study on the Efficacy and Safety of the Combination of Limertinib and Bevacizumab Versus Limertinib Monotherapy as First - Line Treatment for Locally Advanced or Recurrent Metastatic Non - Squamous NSCLC With EGFR Mutations and High PD-L1 Expression.
Brief Title: A Clinical Study on the Efficacy and Safety of the Combination of Limertinib and Bevacizumab Versus Limertinib as First-line Treatment for NSCLC.
Acronym: LIBRA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Zhong Runbo, The chief physician of pneumology department, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-31-25-032614
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: EGFR Mutation Positive Advanced Non Small Cell Lung Cancer; PD-L1 Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Limertinib+bevacizumab
- Control Group (Placebo Comparator)
  Interventions: Drug: Limertinib

INTERVENTIONS:
Drug: Limertinib+bevacizumab — The advanced or metastatic non-small cell lung cancer patients with EGFR mutation and high PD-L1 expression will receive the combination of Limertinib with bevacizuma in first-line treatment
  Other Names: ASK120067
  Arms: Experimental group
Drug: Limertinib — The advanced or metastatic non-small cell lung cancer patients with EGFR mutation and high PD-L1 expression will receive Limertinib in first-line treatment
  Arms: Control Group

SUMMARY:
A prospective, controlled Phase II clinical study on the efficacy and safety of the combination of limertinib and bevacizumab versus limertinib monotherapy as first - line treatment for locally advanced or recurrent metastatic non - squamous NSCLC with EGFR mutations and high PD-L1 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any study - related procedures.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed non - squamous non - small cell lung cancer (NSCLC).
4. Patients with locally advanced (IIIB - IIIC), metastatic, or recurrent (Stage IV) disease, as staged according to the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer (AJCC) 9th edition TNM staging for lung cancer, who are not candidates for surgical or radiation therapy.
5. Confirmed EGFR - sensitive mutations (Ex19del, L858R) in tumor histology or cytology or in hematology.
6. PD - L1 expression with a Combined Positive Score (CPS) ≥ 25%.
7. ECOG performance status score of 0 - 1.
8. No prior treatment with anti - angiogenic inhibitors or EGFR - TKIs.
9. At least one radiologically measurable lesion, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Lesions within a previously irradiated field may be considered measurable if progression has been confirmed.
10. Asymptomatic or symptomatic - stable brain metastases after local treatment are allowed, provided that the following conditions are met: - Measurable disease outside the central nervous system (CNS). - No CNS symptoms or worsening of symptoms within the past 2 weeks. - No need for glucocorticoid treatment, or glucocorticoid treatment discontinued within 7 days prior to the first dose, or stable and reduced glucocorticoid dose to ≤ 10 mg/day prednisone (or equivalent) within 7 days prior to the first dose.
11. Expected survival time > 3 months.
12. Adequate organ function, with the following laboratory values met by subjects: - Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L without the use of granulocyte - colony stimulating factor (G - CSF) within the past 14 days. - Platelets ≥ 100×10⁹/L without blood transfusion within the past 14 days. - Hemoglobin > 9 g/dL without blood transfusion or use of erythropoiesis - stimulating agents within the past 14 days. - Total bilirubin ≤ 1.5× the upper limit of normal (ULN). - Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN (for subjects with liver metastases, ALT or AST ≤ 5×ULN is allowed). - Serum creatinine ≤ 1.5×ULN and creatinine clearance (calculated using the Cockcroft - Gault formula) ≥ 60 ml/min. - Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5×ULN. - Normal thyroid function, defined as thyroid - stimulating hormone (TSH) within the normal range. Subjects may also be included if their baseline TSH is outside the normal range but their total T3 (or free T3) and free T4 are within the normal range. - Cardiac enzyme profile within the normal range (isolated laboratory abnormalities deemed not clinically significant by the investigator are also allowed).
13. For women of childbearing age, a negative urine or serum pregnancy test must be conducted within 3 days prior to the first dose of the study drug (Day 1 of Cycle 1). If the urine pregnancy test result is inconclusive, a blood pregnancy test is required. Non - childbearing - age women are defined as those who have been post - menopausal for at least 1 year, or have undergone surgical sterilization or hysterectomy.
14. All subjects (regardless of gender) with the potential for conception must use contraceptive measures with a failure rate of less than 1% throughout the entire treatment period and until 120 days (or 180 days) after the last dose of the study drug.

Exclusion Criteria:

1. Pathologically diagnosed with small cell lung cancer (SCLC), including lung cancer with a mixture of SCLC and NSCLC.
2. Patients who have received any EGFR - TKI treatment or anti - angiogenic therapy.
3. Received the following treatments: - Systemic anti - tumor treatment such as chemotherapy, targeted therapy, or immunotherapy (including traditional Chinese medicine for anti - tumor purposes) within 3 weeks prior to treatment. - Any investigational drug treatment within 4 weeks prior to treatment. - High - dose immunosuppressive drugs (systemic glucocorticoids exceeding 10 mg/day prednisone or equivalent doses) within 4 weeks prior to treatment. - Attenuated live vaccines within 4 weeks prior to treatment (or planned to receive attenuated live vaccines during the study period). - Major surgery (such as open - cavity, open - chest, or laparotomy) within 4 weeks prior to treatment, or unresolved surgical wounds, ulcers, or fractures.
4. Clinically uncontrollable pleural effusion/peritoneal effusion (subjects who do not require drainage of effusion or whose effusion does not significantly increase after stopping drainage for 3 days are eligible for inclusion).
5. Subjects who received chest radiotherapy with a dose greater than 30Gy within 6 months prior to treatment, or palliative radiotherapy with a dose of 30Gy or less within 7 days prior to treatment (palliative radiotherapy for bone lesions or intracranial lesions is allowed).
6. Active autoimmune diseases that required systemic treatment (such as disease - modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose of study drug. Replacement therapies (such as thyroid hormone, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatment.
7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
8. Known allergy to the active ingredients or excipients of the study drugs bevacizumab and lerotinib.
9. Not fully recovered from the toxicity and/or complications caused by any intervention prior to the start of treatment (i.e., ≤ grade 1 or returned to baseline, excluding fatigue or hair loss).
10. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibodies).
11. Untreated active hepatitis B (defined as positive for HBsAg and HBV - DNA copies greater than the upper limit of normal in the laboratory of the research center). Note: Subjects with hepatitis B who meet the following criteria are also eligible for inclusion: - HBV viral load < 1000 copies/ml (200 IU/ml) prior to the first dose of study drug, and subjects should receive anti - HBV treatment throughout the study drug treatment period to prevent viral reactivation. - For subjects with positive anti - HBc, negative HBsAg, negative anti - HBs, and negative HBV viral load, preventive anti - HBV treatment is not required, but close monitoring for viral reactivation is necessary.
12. Subjects with active HCV infection (positive for HCV antibodies and HCV - RNA levels above the lower limit of detection).
13. Received live vaccines within 30 days prior to the first dose of study drug (Day 1 of Cycle 1). Note: It is allowed to receive injectable inactivated virus vaccines for seasonal influenza within 30 days prior to the first dose of study drug 2: however, intranasal attenuated live influenza vaccines are not allowed. 14. Pregnant or lactating women.

15. Any severe or uncontrolled systemic disease, such as: - Significant and symptomatic abnormalities in rhythm, conduction, or morphology on resting electrocardiogram that are difficult to control, such as complete left bundle branch block, second - degree or higher cardiac conduction block, ventricular arrhythmias, or atrial fibrillation. - Unstable angina, congestive heart failure, chronic heart failure with a New York Heart Association (NYHA) classification of ≥ Grade 2. - Myocardial infarction within 6 months prior to enrollment. - Poorly controlled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg). - History of non - infectious pneumonia that required glucocorticoid treatment within 1 year prior to the first dose of study drug, or current clinically active interstitial lung disease. - Active pulmonary tuberculosis. - Active or uncontrolled infections that require systemic treatment. - Clinically active diverticulitis, intra - abdominal abscess, or gastrointestinal obstruction. - Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis. - Poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L). - Urine routine test indicating proteinuria ≥ ++, and confirmed 24 - hour urine protein quantification > 1.0 g. - Subjects with mental disorders who are unable to cooperate with treatment.

16. Any medical history or evidence of disease, treatment, or laboratory test abnormalities that may interfere with the study results or prevent the subject from fully participating in the study, or other situations deemed by the investigator as unsuitable for inclusion. The investigator considers there are other potential risks that make the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | About 2 years
  the investigator assessed PFS

SECONDARY OUTCOMES:
ORR | about 6 month
  the investigator assessed objective response rate
OS | About 2 years

IPD SHARING:
Plan to Share IPD: Undecided